CLINICAL TRIAL: NCT05298423
Title: Open-label Phase 3 Study of MK-7684A (Coformulation of Vibostolimab With Pembrolizumab) in Combination With Concurrent Chemoradiotherapy Followed by MK-7684A Versus Concurrent Chemoradiotherapy Followed by Durvalumab in Participants With Unresectable, Locally Advanced, Stage III NSCLC
Brief Title: Study of Pembrolizumab/Vibostolimab (MK-7684A) in Combination With Concurrent Chemoradiotherapy Followed by Pembrolizumab/Vibostolimab Versus Concurrent Chemoradiotherapy Followed by Durvalumab in Participants With Stage III Non-small Cell Lung Cancer (MK-7684A-006)
Acronym: KEYVIBE-006
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 7684A-006; MK-7684A-006 (Other: MSD); KEYVIBE-006 (Other: MSD); jRCT2021220015 (Registry Identifier: jRCT); PHRR230831-006071 (Registry Identifier: PHRR); 2022-502752-31-00 (Registry Identifier: EU CT); U1111-1285-3656 (Registry Identifier: UTN); 2021-005135-23 (EudraCT Number)
Record Dates: First submitted 2022-03-17; First posted 2022-03-28 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Cell Death 1 Ligand 1 (PDL1, PD-L1)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; durvalumab; Cisplatin; Pemetrexed; Etoposide; Carboplatin; Paclitaxel

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- pembrolizumab/vibostolimab coformulation+chemotherapy+radiotherapy (Experimental): For the first 3 cycles, participants receive pembrolizumab/vibostolimab (coformulation of 200 mg pembrolizumab and 200 mg vibostolimab) intravenously (IV) on Day 1 plus 3 cycles of investigator's choice of platinum doublet chemotherapy and concurrent standard thoracic radiotherapy during Cycles 2, 3. Participants receive pembrolizumab/vibostolimab for Cycles 4-20 or until discontinuation (up to ~14 months). Cycles 1-20 are 21-day cycles.
  As of protocol amendment 4, participants receiving pembrolizumab/vibostolimab must stop ongoing treatment with pembrolizumab/vibostolimab and will be offered the option to transition to post-cCRT durvalumab consolidation therapy, to complete up to 1 year of consolidation immunotherapy.
  Interventions: Biological: pembrolizumab/vibostolimab; Biological: durvalumab; Drug: cisplatin; Drug: pemetrexed; Drug: etoposide; Drug: carboplatin; Drug: paclitaxel; Radiation: thoracic radiotherapy
- chemotherapy+radiotherapy+durvalumab (Active Comparator): For the first 3 cycles, participants will receive investigator's choice of platinum doublet chemotherapy and concurrent standard thoracic radiotherapy during Cycles 2 and 3. Following concurrent chemoradiotherapy (cCRT), participants receive durvalumab 10 mg/kg every 2 weeks for up to an additional 26 cycles or until discontinuation (up to approximately 14 months). cCRT Cycles 1-3=21-day cycles; durvalumab Cycles 1-26=14-day cycles.
  Interventions: Biological: durvalumab; Drug: cisplatin; Drug: pemetrexed; Drug: etoposide; Drug: carboplatin; Drug: paclitaxel; Radiation: thoracic radiotherapy

INTERVENTIONS:
Biological: pembrolizumab/vibostolimab — Administered as an intravenous (IV) infusion
  Other Names: MK-7684A
  Arms: pembrolizumab/vibostolimab coformulation+chemotherapy+radiotherapy
Biological: durvalumab — Administered as an IV infusion
  Other Names: IMFINZI®
Drug: cisplatin — Cisplatin 75 mg/m^2 administered as an IV infusion in combination with pemetrexed on Day 1 of Cycles 1-3 for non-squamous histology only; In combination with etoposide, cisplatin 50 mg/m^2 is administered on Days 1, 8 of Cycles 1-2 and Days 8, 15 of Cycle 3
  Other Names: PLATINOL-AQ®
Drug: pemetrexed — Pemetrexed 500 mg/m^2 administered as an IV infusion on Day 1 of Cycles 1-3 for non-squamous histology only
  Other Names: ALIMTA®
Drug: etoposide — Etoposide 50 mg/m^2 is administered as an IV infusion on Days 1-5 of Cycles 1-2 and Days 8-12 of Cycle 3;
  Other Names: TOPOSAR®
Drug: carboplatin — Carboplatin area under the curve (AUC) 6 mg/ml/min on Day 1 of Cycle 1 and AUC 2 mg/ml/min on Days 1, 8, 15 of Cycles 2-3, administered as an IV infusion
  Other Names: PARAPLATIN®
Drug: paclitaxel — Paclitaxel 200 mg/m^2 on Day 1 of Cycle 1 and 45 mg/m^2 on Days 1, 8, 15 of Cycles 2-3, administered as an IV infusion
  Other Names: TAXOL®
Radiation: thoracic radiotherapy — 60 Gray [Gy] in 2 Gy fractions for 30 days total administered as an external beam radiation

SUMMARY:
Researchers are looking for new ways to treat people with locally advanced non-small cell lung cancer (NSCLC). The goal of this study is to learn if people who receive the combination of vibostolimab and pembrolizumab (MK-7684A) live longer without the cancer getting worse and live longer overall than people who receive durvalumab.

DETAILED DESCRIPTION:
As of protocol amendment 4, participants receiving combination vibostolimab and pembrolizumab (MK-7684A) discontinued treatment due to lack of efficacy observed in other MK-7684A studies, and are given the option to transition to durvalumab therapy.

ELIGIBILITY:
The main inclusion and exclusion criteria include but are not limited to the following:

Inclusion Criteria

* Has pathologically (histologically or cytologically) confirmed diagnosis of NSCLC.
* Has Stage IIIA, IIIB, or IIIC NSCLC by American Joint Committee on Cancer Version 8
* Is determined to have unresectable, Stage III NSCLC as documented by a multidisciplinary tumor board or by the treating physician in consultation with a thoracic surgeon
* Has no evidence of metastatic disease, indicating Stage IV NSCLC, in whole-body fluorodeoxyglucose (FDG)-positron emission tomography (PET) or FDG-PET/ computed tomography (CT) and CT or magnetic resonance imaging (MRI) scans of diagnostic quality of chest, abdomen, pelvis and brain
* Has measurable disease as defined by RECIST 1.1, with at least 1 lesion being appropriate for selection as a target lesion, as determined by local site investigator/radiology review
* Has not received prior treatment (chemotherapy, targeted therapy, or radiotherapy) for their Stage III NSCLC
* Has provided tumor tissue sample (tissue biopsy [core, incisional, or excisional])
* Has an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1 assessed within 7 days prior to the first administration of study intervention
* Has a life expectancy of at least 6 months

Exclusion Criteria

* Has small cell lung cancer (SCLC) or tumors with the presence of small cell elements. Mixed squamous/nonsquamous tumors are eligible
* Has received prior radiotherapy to the thorax, including radiotherapy to the esophagus, mediastinum, or for breast cancer
* Has received major surgery (with the exception of replacement of vascular access) within 4 weeks before randomization. If the participant had a major operation, the participant must have recovered adequately from the procedure and/or any complications from the operation before starting study intervention
* Is expected to require any other form of antineoplastic therapy, while on study
* Has received colony-stimulating factors (e.g., Granulocyte Colony-Stimulating Factor [G-CSF], Granulocyte Macrophage Colony-Stimulating Factor [GM-CSF], or recombinant erythropoietin) within 28 days prior to the first dose of study intervention
* Has received a live or live-attenuated vaccine within 30 days before the first dose of study intervention
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks before the first dose of study intervention
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study medication
* Has a known additional malignancy that is progressing or has required active treatment within the past 5 years
* Has an active autoimmune disease that has required systemic treatment in past 2 years
* Has a history of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Has an active infection requiring systemic therapy
* Has a known history of human immunodeficiency virus (HIV) infection
* Has a known history of Hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV ribonucleic acid [RNA] qualitative is detected) infection
* Has had an allogenic tissue/solid organ transplant

Pemetrexed-specific Criteria:

* Is unable to interrupt aspirin or other nonsteroidal anti-inflammatory drugs (NSAIDs), other than an aspirin dose ≤1.3 grams per day, for at least 2 days (5 days for long-acting agents [for example, piroxicam]) before, during, and for at least 2 days after administration of pemetrexed
* Is unable/unwilling to take folic acid, vitamin B12, and dexamethasone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 611 (Actual)
Dates: Start 2022-05-03 (Actual); Primary Completion 2026-08-19 (Estimated); Study Completion 2026-08-19 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Who Experience at Least One Adverse Event (AE) | Up to approximately 48 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Number of Participants Who Discontinue Study Treatment Due to an Adverse Event (AE) | Up to approximately 48 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (160):
- United States (21):
  - VA Long Beach Healthcare System ( Site 2831), Long Beach, California
  - VA West Los Angeles Medical Center ( Site 2808), Los Angeles, California
  - Millennium Oncology Research Clinic ( Site 2801), Hollywood, Florida
  - Mid Florida Hematology and Oncology Center ( Site 2800), Orange City, Florida
  - Moffitt Cancer Center ( Site 2818), Tampa, Florida
  - University of Chicago Medical Center ( Site 2828), Chicago, Illinois
  - Franciscan St. Francis Health ( Site 2812), Indianapolis, Indiana
  - MFSMC-HJWCI ( Site 2804), Baltimore, Maryland
  - Boston Medical Center ( Site 2829), Boston, Massachusetts
  - University of Massachusetts Chan Medical School ( Site 2815), Worcester, Massachusetts
  - University of Missouri Hospital ( Site 2839), Columbia, Missouri
  - Cox Medical Center North-Cox Medical Center/Hulston Cancer Center/ Radiation Oncology ( Site 2837), Springfield, Missouri
  - Rutgers Cancer Institute of New Jersey ( Site 2805), New Brunswick, New Jersey
  - Icahn School of Medicine at Mount Sinai ( Site 2821), New York, New York
  - White Plains Hospital ( Site 2835), White Plains, New York
  - Kaiser Permanente Northwest-Central Interstate--Oncology ( Site 2816), Portland, Oregon
  - Lancaster General Hospital - Ann B Barshinger Cancer Institute ( Site 2827), Lancaster, Pennsylvania
  - Thomas Jefferson University - Clinical Research Institute ( Site 2813), Philadelphia, Pennsylvania
  - Millennium Research & Clinical Development ( Site 2811), Houston, Texas
  - Central Texas Veterans health care-Oncology & Hematology ( Site 2819), Temple, Texas
  - MultiCare Health System ( Site 2817), Tacoma, Washington
- Argentina (3):
  - Clinica Adventista Belgrano ( Site 3601), Caba., Buenos Aires F.D.
  - Instituto Médico Río Cuarto ( Site 3600), Río Cuarto, Córdoba Province
  - Sanatorio Parque ( Site 3602), Rosario, Santa Fe Province
- Australia (5):
  - Canberra Hospital ( Site 0010), Canberra, Australian Capital Territory
  - Icon Cancer Centre Hobart ( Site 0003), Hobart, Tasmania
  - Ballarat Health Services-Medical Oncology ( Site 0002), Ballarat Central, Victoria
  - Frankston Hospital-Oncology and Haematology ( Site 0009), Frankston, Victoria
  - St Vincent's Hospital-Oncology Clinical Trials ( Site 0005), Melbourne, Victoria
- Brazil (3):
  - Hospital Nossa Senhora da Conceição ( Site 0111), Porto Alegre, Rio Grande do Sul
  - Instituto de Educação, Pesquisa e Gestão em Saúde ( Site 0105), Rio de Janeiro
  - A. C. Camargo Cancer Center-CAPEC ( Site 0102), São Paulo
- Chile (6):
  - FALP-UIDO ( Site 0205), Santiago, Region M. de Santiago
  - Centro de Oncología de Precisión ( Site 0209), Santiago, Region M. de Santiago
  - Bradfordhill ( Site 0200), Santiago, Region M. de Santiago
  - James Lind Centro de Investigacion del Cancer ( Site 0202), Temuco, Región de la Araucanía
  - ONCOCENTRO APYS-ACEREY ( Site 0203), Viña del Mar, Región de Valparaíso
  - Biocenter ( Site 0208), Concepción, Región del Biobío
- China (28):
  - Beijing Cancer hospital-intrathoratic deparmtment II ( Site 0328), Beijing, Beijing Municipality
  - Beijing Cancer hospital-Oncology Radiotherapy Department ( Site 0309), Beijing, Beijing Municipality
  - Beijing Peking Union Medical College Hospital-pneumology department ( Site 0300), Beijing, Beijing Municipality
  - Army Medical Center of People's Liberation Army-Oncology Department ( Site 0321), Chongqing, Chongqing Municipality
  - Fujian Provincial Cancer Hospital ( Site 0316), Fuzhou, Fujian
  - Fujian Medical University Union Hospital-1 Bingfanglou ( Site 0330), Fuzhou Fujian, Fujian
  - The First Affiliated hospital of Xiamen University-oncology ( Site 0317), Xiamen, Fujian
  - Southern Medical University Nanfang Hospital-Department of Oncology ( Site 0336), Guangzhou, Guangdong
  - Fourth Hospital of Hebei Medical University ( Site 0331), Shijiazhuang, Hebei
  - Henan Cancer Hospital ( Site 0333), Zhengzhou, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology ( Site 0315), Wuhan, Hubei
  - Hubei Cancer Hospital ( Site 0311), Wuhan, Hubei
  - Xiangya Hospital Central South University-Oncology department ( Site 0310), Changsha, Hunan
  - Hunan Cancer Hospital ( Site 0307), Changsha, Hunan
  - The Second Affiliated Hospital of Soochow University ( Site 0314), Suzhou, Jiangsu
  - Affiliated Hospital of Jiangsu University ( Site 0305), Zhenjiang, Jiangsu
  - Jilin Cancer Hospital-oncology department ( Site 0319), Changchun, Jilin
  - Shandong Provincial Hospital ( Site 0326), Jinan, Shandong
  - Qingdao Central Hospital-Endocrinology ( Site 0332), Qingdao, Shandong
  - Shanghai Chest Hospital-Radiotherapy Department ( Site 0306), Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center ( Site 0304), Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital-Radiotherapy department ( Site 0335), Shanghai, Shanghai Municipality
  - Shanxi Cancer Hospital-Pulmonology ( Site 0322), Taiyuan, Shanxi
  - West China Hospital of Sichuan University ( Site 0324), Chengdu, Sichuan
  - Tianjin Cancer Hospital ( Site 0329), Tianjin, Tianjin Municipality
  - Hangzhou Cancer Hospital-Medical Oncology ( Site 0302), Hangzhou, Zhejiang
  - The Second Affiliated hospital of Zhejiang University school of medicine ( Site 0301), Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital ( Site 0308), Hangzhou, Zhejiang
- Costa Rica (3):
  - CIMCA ( Site 0501), San José, Provincia de San José
  - PROCLINICAL Pharma ( Site 0504), San José, Provincia de San José
  - Hospital Metropolitano - Sede Lindora ( Site 0503), Santa Ana, Provincia de San José
- Czechia (2):
  - Masarykuv onkologicky ustav ( Site 3500), Brno, Brno-mesto
  - Fakultni nemocnice Ostrava-Klinika onkologicka ( Site 3502), Ostrava, Moravskoslezský kraj
- Dominican Republic (2):
  - Instituto de Oncologia ( Site 3003), Santo Domingo, Nacional
  - Onconet ( Site 3002), Distrito Nacional, Santo Domingo Province
- Germany (4):
  - Klinikum Chemnitz-Klinik für Innere Medizin IV ( Site 0607), Chemnitz, Saxony
  - LungenClinic Grosshansdorf-Onkologie ( Site 0602), Großhansdorf, Schleswig-Holstein
  - Universitaetsklinikum Schleswig-Holstein Campus Kiel-Medizinische Klinik II, Hämatologie und Onkolo ( Site 0609), Kiel, Schleswig-Holstein
  - Charité Campus Virchow-Klinikum-Department of Infectious Diseases and Pulmonary Medicine ( Site 0603), Berlin
- Greece (7):
  - Errikos Dunant Hospital Center-Second Department of Oncology and Clinical Trials Unit ( Site 0703), Athens, Attica
  - Alexandra General Hospital of Athens-ONCOLOGY DEPT. ( Site 0706), Athens, Attica
  - Sotiria Thoracic Diseases Hospital of Athens ( Site 0704), Athens, Attica
  - Metropolitan Hospital ( Site 0702), Athens, Attica
  - General Oncology Hospital of Kifissia "Agioi Anargiroi"-2nd Department of Medical Oncology ( Site 0705), Nea Kifissia, Attica
  - University General Hospital of Heraklion-Internal Medicine-Oncology ( Site 0700), Heraklion, Irakleio
  - European Interbalkan Medical Center ( Site 0701), Thessaloniki
- Guatemala (4):
  - MEDI-K ( Site 0807), Guatemala City
  - Private Practice- Dr. Rixci Augusto Lenin Ramírez ( Site 0802), Guatemala City
  - Centro Regional de Sub Especialidades Médicas SA ( Site 0801), Quetzaltenango
  - Centro Medico Integral De Cancerología (CEMIC) ( Site 0805), Quetzaltenango
- Israel (5):
  - Rambam Health Care Campus-Oncology ( Site 1001), Haifa
  - Shaare Zedek Medical Center ( Site 1003), Jerusalem
  - Rabin Medical Center ( Site 1004), Petah Tikva
  - Sheba Medical Center-ONCOLOGY ( Site 1000), Ramat Gan
  - Sourasky Medical Center ( Site 1002), Tel Aviv
- Italy (7):
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale-Oncologia medica Toraco-Polmonare ( Site 1107), Napoli, Campania
  - Policlinico Universitario Campus Bio-Medico-Radiation Oncology ( Site 1101), Rome, Lazio
  - Fondazione IRCCS Istituto Nazionale dei Tumori ( Site 1100), Milan, Lombardy
  - Ospedale San Gerardo-ASST Monza-Oncologia ( Site 1102), Monza, Lombardy
  - Azienda Ospedaliera Spedali Civili di Brescia ( Site 1105), Brescia
  - Ospedale San Raffaele. ( Site 1104), Milan
  - Fondazione IRCCS Policlinico San Matteo ( Site 1103), Pavia
- Japan (13):
  - National Hospital Organization Shikoku Cancer Center ( Site 1211), Matsuyama, Ehime
  - Kurume University Hospital ( Site 1212), Kurume, Fukuoka
  - Kobe Minimally Invasive Cancer Center ( Site 1210), Kobe, Hyōgo
  - Kanagawa Cancer Center ( Site 1204), Yokohama, Kanagawa
  - Miyagi Cancer Center ( Site 1200), Natori-shi, Miyagi
  - Sendai Kousei Hospital ( Site 1213), Sendai, Miyagi
  - Niigata Cancer Center Hospital ( Site 1205), Niigata, Niigata
  - Kansai Medical University Hospital ( Site 1207), Hirakata, Osaka
  - Osaka Medical and Pharmaceutical University Hospital ( Site 1208), Takatsuki, Osaka
  - Saitama Prefectural Cancer Center ( Site 1201), Ina-machi, Saitama
  - Cancer Institute Hospital of JFCR ( Site 1202), Koto, Tokyo
  - Showa Medical University Hospital ( Site 1203), Shinagawa, Tokyo
  - Osaka International Cancer Institute ( Site 1209), Osaka
- Malaysia (3):
  - University Malaya Medical Centre-Clinical Oncology ( Site 1402), Lembah Pantai, Kuala Lumpur
  - Hospital Pulau Pinang ( Site 1400), George Town, Pulau Pinang
  - Hospital Kuala Lumpur-Radiotherapy and Oncology ( Site 1401), Kuala Lumpur
- Mexico (4):
  - Actualidad Basada en la Investigación del Cáncer-Lung Cancer ( Site 1505), Guadalajara, Jalisco
  - Arké SMO S.A. de C.V. ( Site 1504), Mexico City, Mexico City
  - Centro Oncologico de Chihuahua-Unidad de Investigacion Clinica ( Site 1507), Chihuahua City
  - Centro de Investigacion Clinica de Oaxaca ( Site 1501), Oaxaca City
- Philippines (2):
  - THE MEDICAL CITY-Cancer Research Center ( Site 3200), Pasig, National Capital Region
  - Veterans Memorial Medical Center-Section of Oncology ( Site 3201), Quezon City, National Capital Region
- Portugal (4):
  - Champalimaud Foundation ( Site 2003), Lisbon, Lisbon District
  - Hospital CUF Descobertas ( Site 2006), Lisbon, Lisbon District
  - Unidade Local de Saude de Santo António - Hospital Santo António ( Site 2004), Porto
  - Instituto Português de Oncologia do Porto Francisco Gentil, EPE ( Site 2001), Porto
- Romania (6):
  - Centrul Medical Medicover Victoria ( Site 2106), Bucharest, București
  - Amethyst Radiotherapy Center ( Site 2102), Florești, Cluj
  - Centrul de Oncologie "Sfântul Nectarie" ( Site 2100), Craiova, Dolj
  - Radiology Therapeutic Center ( Site 2108), Otopeni, Ilfov
  - Cabinet Medical Oncomed ( Site 2101), Timișoara, Timiș County
  - Centrul Medical Neolife- Baneasa ( Site 2110), Bucharest
- South Africa (5):
  - CANCERCARE LANGENHOVEN DRIVE ONCOLOGY CENTRE ( Site 2304), Port Elizabeth, Eastern Cape
  - Wilgers Oncology Centre ( Site 2301), Pretoria, Gauteng
  - The Oncology Centre ( Site 2300), Durban, KwaZulu-Natal
  - Abraham Oncology ( Site 2303), Richards Bay, KwaZulu-Natal
  - Cape Town Oncology Trials ( Site 2306), Cape Town, Western Cape
- South Korea (4):
  - The Catholic University Of Korea St. Vincent's Hospital-Medical Oncology ( Site 2401), Suwon, Kyonggi-do
  - Ajou University Hospital-Hematology-Oncology ( Site 2402), Suwon, Kyonggi-do
  - Chungbuk National University Hospital-Internal medicine ( Site 2400), Cheongju-si, North Chungcheong
  - Severance Hospital, Yonsei University Health System-Lung Cancer Center ( Site 2403), Seoul
- Spain (4):
  - Hospital Universitari Vall d'Hebron ( Site 2501), Barcelona, Catalonia
  - HOSPITAL CLÍNIC DE BARCELONA-ICHMO- Clinic Institut of Haematological and Oncological diseases ( Site 2503), Barcelona, Catalonia
  - CHUS - Hospital Clinico Universitario-Servicio de Oncologia ( Site 2502), Santiago de Compostela, La Coruna
  - HOSPITAL UNIVERSITARIO QUIRONSALUD MADRID-ONCOLOGIA MEDICA ( Site 2504), Pozuelo de Alarcón, Madrid, Comunidad de
- Turkey (Türkiye) (9):
  - Medipol Mega Universite Hastanesi-oncology ( Site 2611), Stanbul, Istanbul
  - Ege University Medicine of Faculty-Chest Diseases Department ( Site 2603), Bornova, İzmir
  - Baskent University Dr. Turgut Noyan Research and Training Center-ONCOLOGY ( Site 2607), Adana
  - Ankara Gülhane Eitim ve Aratrma Hastanesi-Oncology ( Site 2602), Ankara
  - Hacettepe Universitesi-oncology hospital ( Site 2605), Ankara
  - Memorial Ankara Hastanesi-Medical Oncology ( Site 2609), Ankara
  - Ankara City Hospital-Medical Oncology ( Site 2601), Ankara
  - TC Saglik Bakanligi Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi-oncology ( Site 2610), Istanbul
  - I.E.U. Medical Point Hastanesi-Oncology ( Site 2612), Izmir
- Ukraine (6):
  - Limited Liability Company Ukrainian Center of Tomotherapy-Department of Chemotherapy ( Site 2905), Kropyvnytskyi, Kirovohrad Oblast
  - Municipal non-profit enterprise "Lviv Territorial Medical Union "Multidisciplinary Clinical Hospital ( Site 2920), Lviv, Lviv Oblast
  - Rivne Regional Clinical Hospital ( Site 2919), Rivne, Rivne Oblast
  - Communal Noncommercial Enterprise "Podillia Regional Oncology Center Of Vinnytsia Regional Council" ( Site 2900), Vinnytsia, Vinnytsia Oblast
  - Volyn Regional clinical hospital. Regional Medical Oncology Centre. Oncology chemotherapy department ( Site 2918), Lutsk, Volyn Oblast
  - Universal Clinic Oberig-Oncology Center ( Site 2916), Kyiv

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26317&tenant=MT_MSD_9011